CLINICAL TRIAL: NCT01793506
Title: Novel Testing Procedures for Detection of Primary Humoral Immunodeficiency
Brief Title: Novel Testing Procedures
Status: Withdrawn | Type: Observational
Why Stopped: Never funded or completed
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Baxter-01; 01 (Other Grant/Funding Number: Baxter)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-01

CONDITIONS: Immunodeficiencies
Keywords: immunodeficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PID: Any subject having testing done to evaluate the immune system is eligible for this study. This will include patients with known PIDs as well as patients evaluated for a suspected immunodeficiency.

SUMMARY:
The purpose of this study is to evaluate a novel screening test to detect patients with primary immunodeficiencies(PIDs). The investigators plan to use information gained from this study in order to advance the field of clinical immunology, thus improving the diagnosis, treatment, and well-being of future patients. The purpose of this study is to determine if this screening test is able to detect patients with immune problems, and the investigators will test patients with known PIDs to determine if the test is accurate

The investigators hypothesize that detecting serum immunoglobulins from dried blood spots will be effective in detecting patients with known primary immunodeficiencies. If our hypothesis is confirmed, it opens the possibility of using point of care testing to screen for primary immune deficiencies.

Age of study subjects will range from 1 year to 80 years of age, and will be recruited form the Immunodeficiency clinic at the Medical College of Wisconsin/Children's Hospital of Wisconsin (MCW/CHW). Any subject having testing done to evaluate the immune system is eligible for this study. This will include patients with known PIDs as well as patients evaluated for a suspected immunodeficiency. It is anticipated that 150 subjects will be analyzed over a two year period.

DETAILED DESCRIPTION:
After consent is obtained, blood will be obtained. The total amount of blood to drawn in one day will not exceed 1.5 mL (1/3 tsp) per pound of body weight. All samples will be collected at the same time as routine blood draws as ordered by your physician.

Subject samples will be de-identified by the Principal Investigator (PI) and given a serial number. The PI will retain a secured log of the serial numbers and basic identifiers (name, Date of Birth (DOB0, sex, preliminary diagnosis, and test results), and the subject samples will be stored in a secured freezer. Only the PI will have access to the secured log book. All study test results will be kept on compact discs, or similar computer storage devices, in a secured area that will only be accessible by the PI. Study test results will not kept on computers accessible by other individuals. The samples will not be sold to any third party. The results of this research will not be conveyed to any third party. If the subject withdraws or is withdrawn from the study all identifiable biological samples from that subject will be discarded. The sample will not be available for any other type of testing outside of this study.

ELIGIBILITY:
Inclusion Criteria:

* Any subject having testing done to evaluate the immune system is eligible for this study.

Exclusion Criteria:

* Inability or unwillingness on the part of the parents or individual to provide clinical or family history, or refusal to allow blood sampling.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female, 1 year to 80 years of age
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clinically validated diagnostic test for primary humoral immunodeficiency. | two years
  We will test if measurement of serum immunoglobulin levels from a blood spot on filter paper is able to detect patients with known immunodeficiencies and low Immunoglobulin G levels.

CONTACTS AND LOCATIONS:
Overall Officials: James Verbsky, MD PhD, Principal Investigator — Medical College of Wisconsin; John Routes, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Asthma, Allergy & Immunology Clinics Medical College of Wisconsin, Milwaukee, Wisconsin, United States